CLINICAL TRIAL: NCT02493569
Title: A Multicenter Study of Clinical Epidemiology of Breast Cancer in Shaanxi Province of China (Based on Hospital)
Brief Title: A Multicenter Study of Clinical Epidemiology of Breast Cancer in Shaanxi Province of China
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Other Study IDs: KYLLSL-2015-153-01
Record Dates: First submitted 2015-07-07; First posted 2015-07-09 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2016-08

CONDITIONS: Breast Cancer
Keywords: Breast cancer, hospital, epidemiology, diagnosis, treatment
MeSH Terms: conditions — Breast Neoplasms; Disease

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Epidemiology breast cancer patients: Observe the features of clinical diagnosis and treatment for female breast cancer patients
  Interventions: Procedure: The radical mastectomy of breast cancer

INTERVENTIONS:
Procedure: The radical mastectomy of breast cancer — The radical mastectomy of breast cancer could be used for the treatment of breast cancer during the observation.

SUMMARY:
The purpose of the study is to study the epidemic features and diagnosis of female breast cancer, especially the diagnosis and treatment of breast cancer.The disease-free survival (DFS) and the total survival time(OS) of the breast cancer patients will also be studied.

DETAILED DESCRIPTION:
The study is a multicentric, retrospective clinical study based on the hospital. The target number of cases are X patients who are eligible for breast cancer after radical mastectomy. To collect the clinicopathological data and treatment data of the breast cancer patients and do the follow-up visit of all the patients who are included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Female patients;
* The hospitalized patients who are confirmed of the primary breast cancer histologically;
* The date of the inpatients are within the month we chosen;
* Patients who are within the month we chosen have been received or under receiving the relevant treatment including surgical treatment, chemotherapy and radiotherapy.

Exclusion Criteria:

* Male breast cancer patients;
* Patients with breast cancer who are not under the chosen time;
* Non hospitalized patients.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The female breast cancer patients in Shaanxi Province of China, those study population shoud be the hospitalized patients who are confirmed of the primary breast cancer histologically, moreover, the date of the inpatients are within the month we chosen and those inpatients should have been received or under receiving the relevant treatment including surgical treatment, chemotherapy and radiotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Overall five-year survival for the female breast cancer patients | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Yu Ren, MD,PhD, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University